CLINICAL TRIAL: NCT03137420
Title: Psychological Distress in Relatives of Severely Injured Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00074
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Polytrauma; Psychological Distress; Relatives
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severely injured patients and their relatives: Severely injured patients (ISS > 16) and their relatives. Relatives are defined as on of the following: spouse/partner, son/daughter, parent, sibling, cousin.
  Interventions: Diagnostic Test: Numeric Scale of Family Distress
- Monotrauma patients and theri relatives: Patients with isolated non-life threatening musculo-skeletal injuries and their relatives (control). Relatives are defined as on of the following: spouse/partner, son/daughter, parent, sibling, cousin.
  Interventions: Diagnostic Test: Numeric Scale of Family Distress

INTERVENTIONS:
Diagnostic Test: Numeric Scale of Family Distress — Questionnaires at 1, 3, 6 and 12 months
  Other Names: Hospital Anxiety and Depression Scale; Brief Family Distress Scale

SUMMARY:
Patients who have sustained and survived a polytrauma do heavily depend on the support and functioning of their family. This is only possible if the family members are physically and mentally able to cope with the situation.

It is the investigators' hypothesis that the true percentage of polytrauma patients' relatives suffering under relevant psychological distress is higher than commonly assumed.

The investigators conduct a prospective cohort study where we follow up on a cohort of patients and their relatives over 1 year after trauma - one group with severely injured patients (case) and one group with minor musculo-skeletal injuries (control).

In order to assess the influence of the patients' disability and their own psychological distress on the psychological distress of the relatives, the investigators also collect corresponding data from the patients themselves.

In order to assess the influence of the trauma itself, the investigators compare a group of multiple injured patients and their relatives with a group of patients with isolated musculoskeletal injuries and their relatives. In addition, the investigators record the ISS of each patient. In order to investigate the changes in relatives' distress over time and to find out more about potential risk factors or con-founders it is necessary to conduct a prospective study.

DETAILED DESCRIPTION:
Background The incidence of polytrauma has been estimated to range between 25 and 52 per 100'000 in Europe. Severely injured patients are known to suffer increased psychological distress and early identification of these patients can help to provide resources and support for coping strategies. The long-term physical and mental health of such polytrauma survivors can be improved by the presence of a supporting network including patients support groups, social support networking, and - most important - family and friends.

While it has been shown that caring for a family member with chronic disease like cancer or disability after isolated traumatic brain injury or a stroke is associated with significant distress for relatives, little is known on how families function and cope after one of them has had an accident with multiple severe injuries.

Rationale for the research project Patients who have sustained and survived a polytrauma do heavily depend on the support and functioning of their family. This is only possible if the family members are physically and mentally able to cope with the situation.

It is the study's hypothesis that the true percentage of polytrauma patients' relatives suffering under relevant psychological distress is higher than commonly assumed. It is the investigators' strong opinion that it would be important to identify these individuals early (e.g. by a screening test as the one developed in this study) in order to help the helpers.

Objectives

Primary objective: to investigate the psychological impact on relatives of having a severely injured patient as family member in dependence of:

* the patient's disability and psychological stress
* the severity of the trauma (multiple injuries vs isolated musculoskeletal injury) Secondary objective: to develop a simple screening test (Numeric Scale of Distress) and to validate it against existing more complex scoring systems.

Primary and secondary endpoint/outcome(s) Primary outcome: Hospital Anxiety and Depression Scale (HADS) at 1, 3, 6 and 12 months Secondary outcomes: Brief Family Distress Scale (BFDS) and Numeric Scale of Family Distress (NSFD) at 1, 3, 6 and 12 months c) Screening test: Correlation between NSFD and HADS, and NSFD and BFDS

Other study variables

* Patient's age and gender
* Patient's pattern of injury (Abbreviated Injury Scale [AIS] & Injury Severity Score [ISS])
* Patient's injury result of interperson-violence [Yes/No]
* Patient's degree of disability (Stanford HAQ 8-Item Disability Scale; HAQDS)
* Patient's situation of living (home no help, home with support, nursing home)
* Relative's age and gender
* Relative's degree of kinship (spouse/partner, son/daughter, parent, sibling, cousin)

Design Prospective study In order to confirm the investigators's primary hypothesis that the true percentage of polytrauma patients' relatives suffering under relevant psychological distress is higher than commonly assumed we follow up on a cohort of patients and their relatives over 1 year after trauma - one group with severely injured patients (case) and one group with minor musculo-skeletal injuries (control).

In order to assess the influence of the patients' disability and their own psychological distress on the psychological distress of the relatives, the investigators also collect corresponding data from the patients themselves.

In order to assess the influence of the trauma itself, the investigators compare a group of multiple injured patients and their relatives with a group of patients with isolated musculoskeletal injuries and their relatives. In addition, the investigators record the ISS of each patient In order to investigate the changes in relatives' distress over time and to find out more about potential risk factors or confounders it is necessary to conduct a prospective study.

Procedures

1. a list of severely injured patients and patients with isolated non-life threatening musculo-skeletal injuries will be generated from the intern Polytrauma Database and the clinical information system. Only those individuals will have access to this data, that had already been involved into the treatment of these patients or otherwise had by law the right to access the charts (in order not to violate the command of professional confidentiality).
2. within 6 weeks of the initial trauma, patients and their relatives who are eligible according to the inclusion and exclusion criteria will be contacted by phone and will be asked if they would be willing to participate (duration for each participant: 5 min, in most cases only the patient or one member of the family will be contacted as a first representative). During this phone call, also the basic ability to understand German language will be assessed.
3. if agreed, the patient and their relatives will be send the study information, the informed consent form and a short questionnaire containing the HADS (14 items), the BFDS (1 item), and the NSFD (1 numeric scale)as well as questions regarding the other variables listed above under 4.3. The questionnaires will be number-coded. The patient will be asked to complete the HAQDS (8 items), in addition. Completion of the whole questionnaire will take about 10 min per participant. The participants will be asked to send back the signed informed consent and the completed questionnaire.
4. if there is no response to step 2 or 3, the participants will be contacted by phone or mail once more
5. the returned questionnaires will be evaluated for presence of informed consent and then transferred into a number-coded REDCap data file. Only the research team will have access to the main data file and only the project leader will have access to the code key. Both files will be stored on a research server of the Klinik für Traumatologie, UniversitätsSpital Zürich.

Criteria for withdrawal / discontinuation of participants

A participant will be discontinued from the project in case of:

* withdrawal of informed consent
* non-compliance In such case, all health-related data that has already been acquired will be anonymized upon termination of data analysis or - if anonymization is not possible - will be kept for further analysis as the patient was informed and gave consent to at the beginning of the project.

ELIGIBILITY:
Inclusion criteria

* age ≥ 18 years
* Severely injured patients and their relatives (ISS > 16) orpatients with isolated non-life threatening musculo-skeletal injuries and their relatives (control). Relatives are defined as on of the following: spouse/partner, son/daughter, parent, sibling, cousin.
* patients admitted to the Klinik für Traumatologie, UniversitätsSpital Zürich, during the years 2017/18 and their relatives (control)

Exclusion criteria

* Patients who are still in a life-threatening situation and their relatives
* Patients and relatives without signed informed consent
* Participants with cognitive disabilities not allowing to complete the questionnaires or to give informed consent (their relatives can still be included as the relatives of disabled patients most likely suffer under pronounced distress)
* Participants that are able to read and understand German language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 prospective severely injured patients and their relatives (cases) and 50 prospective patients with isolated non-life threatening musculo-skeletal injuries and their relatives (control).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Questionnaire on anxiety and depression

SECONDARY OUTCOMES:
Brief Family Distress Scale (BFDS) | 12 months
  Questionnaire on subjective distress in a family
Numeric Scale of Family Distress (NSFD) | 12 months
  Scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Georg Osterhoff, MD, Principal Investigator — University of Zurich
Locations (1):
- Division of Trauma Surgery, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No